CLINICAL TRIAL: NCT01868568
Title: A Randomised, Double-blind, Multiple Period Cross-over Trial Comparing Insulin 454 and Insulin Aspart Fixed Combination Products With Separately Injected, Simultaneous Doses of Insulin 454 and Insulin Aspart, Compared to Biphasic Insulin Aspart 30 (NovoMix® 30) in Subjects With Type 1 Diabetes
Brief Title: Comparison of IDegAsp (Inclusive Three Explorative Formulations) With Insulin Degludec and Insulin Aspart Separately Injected in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1959; 2007-006110-42 (EudraCT Number)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- IDegAsp 30 + placebo (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 30; Drug: placebo
- Insulin aspart + insulin degludec - low concentration 1 (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IDegAsp 40 + placebo (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 40; Drug: placebo
- Insulin aspart + insulin degludec - high concentration 1 (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IDegAsp 45 + placebo (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 45; Drug: placebo
- Insulin aspart + insulin degludec (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IDegAsp 55 + placebo (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 55; Drug: placebo
- Insulin aspart + insulin degludec - high concentration (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- BIAsp 30 + placebo (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: placebo

INTERVENTIONS:
Drug: insulin degludec — Administered subcutaneously (s.c., under the skin).
  Arms: Insulin aspart + insulin degludec; Insulin aspart + insulin degludec - high concentration; Insulin aspart + insulin degludec - high concentration 1; Insulin aspart + insulin degludec - low concentration 1
Drug: insulin degludec/insulin aspart 30 — A single dose administered subcutaneously (s.c., under the skin).
  Arms: IDegAsp 30 + placebo
Drug: insulin degludec/insulin aspart 40 — A single dose administered subcutaneously (s.c., under the skin).
  Arms: IDegAsp 40 + placebo
Drug: insulin degludec/insulin aspart 45 — A single dose administered subcutaneously (s.c., under the skin).
  Arms: IDegAsp 45 + placebo
Drug: insulin degludec/insulin aspart 55 — A single dose administered subcutaneously (s.c., under the skin).
  Arms: IDegAsp 55 + placebo
Drug: insulin aspart — A single dose administered subcutaneously (s.c., under the skin).
  Arms: Insulin aspart + insulin degludec; Insulin aspart + insulin degludec - high concentration; Insulin aspart + insulin degludec - high concentration 1; Insulin aspart + insulin degludec - low concentration 1
Drug: biphasic insulin aspart 30 — A single dose administered subcutaneously (s.c., under the skin).
  Arms: BIAsp 30 + placebo
Drug: placebo — A single dose administered subcutaneously (s.c., under the skin).
  Arms: BIAsp 30 + placebo; IDegAsp 30 + placebo; IDegAsp 40 + placebo; IDegAsp 45 + placebo; IDegAsp 55 + placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare insulin degludec and insulin aspart (IDegAsp) co-formulations with separately injected, simultaneous doses of insulin degludec (insulin 454) and insulin aspart, compared with biphasic insulin aspart 30 (NovoMix® 30) in subjects with type 1 diabetes mellitus. Each subject will be randomised to four out of nine possible treatment arms. IDegAsp 40, IDegAsp 45, IDegAsp 55 and IDeg high concentration were explorative formulations, not similar to the proposed commercial formulation.

ELIGIBILITY:
Inclusion Criteria:

* Glycosylated haemoglobin A1c (HbA1c) below or equal to 10.0 % based on central laboratory results
* Diagnosed with type 1 diabetes and treated with insulin for above or equal to 12 months
* Body Mass Index (BMI) between 18.0 and 27.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* A subject with a history of significant multiple drug allergies or with a known or suspected allergy to the trial product or any medicine chemically related to the trialproduct, as judged by the Investigator
* A subject who is known to have hepatitis or who is carrier of the Hepatitis B surface antibodies, or has a positive result to the test for HIV antigen (HBsAg) or Hepatitis C antibodies
* A subject who has participated in any other trials involving investigational products within the 3 months preceding the start of dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart concentration curve | 0-2 hours after dosing

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve | 0-26 hours after dosing
Area under the serum insulin 454 concentration curve | 0-120 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com